CLINICAL TRIAL: NCT01016262
Title: A Multicenter, Double-blind, Controlled, Randomized, Parallel Group Comparison Phase IIIa Treatment Investigation on the Efficacy and Safety of MAX-002 Suppository Versus Placebo and Active Medicine in Mild to Moderate Ulcerative Proctitis
Brief Title: Efficacy and Safety Study of MAX-002 Suppository Versus Placebo and Active Medicine in Mild to Moderate Ulcerative Proctitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision was taken solely for business/administrative reasons, no safety considerations entered into this. Ongoing randomized patients to complete.
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-ME-CAPSITUP508-01
Record Dates: First submitted 2009-11-17; First posted 2009-11-19 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Proctitis, Ulcerative
Keywords: Ulcerative proctitis; Proctocolitis; Inflammatory Bowel Disease; Gastrointestinal Diseases; Colonic Diseases; Mesalamine; 5-ASA
MeSH Terms: conditions — Proctitis; Ulcer; Proctocolitis; Inflammatory Bowel Diseases; Gastrointestinal Diseases; Colonic Diseases | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MAX-002 (Experimental)
  Interventions: Drug: MAX-002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Canasa® (Active Comparator)
  Interventions: Drug: Canasa®

INTERVENTIONS:
Drug: MAX-002 — MAX-002 suppository 1 gram (g) rectally once daily at bedtime for 6 weeks during the DB phase. Participants will then receive either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the open-label (OL) phase.
  Other Names: Mesalamine
  Arms: MAX-002
Drug: Placebo — Matching placebo suppository rectally once daily at bedtime for 6 weeks during the DB phase. Participants will then receive either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
  Arms: Placebo
Drug: Canasa® — Canasa® suppository 1 g rectally once daily at bedtime for 6 weeks during the DB phase. Participants will then receive either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
  Other Names: Mesalamine
  Arms: Canasa®

SUMMARY:
This is a prospective, multicenter, double-blind (DB), controlled, randomized, parallel group comparison Phase 3a study to evaluate the efficacy and safety of new mesalamine suppositories (MAX-002) as compared to placebo and active medicine after 6 weeks of treatment in adults with mild to moderate ulcerative proctitis (UP).

DETAILED DESCRIPTION:
The present study consists of screening period (2 weeks before randomization), DB phase (6 weeks), OL phase (8 weeks) and follow-up visits at Week 3, Week 6 and Week 14. Participants who are eligible will be randomized to receive 1g MAX-002, 1g Canasa® and placebo suppository once daily in the DB phase. Participants who complete or discontinue the study at Week 6 will either receive 1g MAX-002 suppositories on a voluntary basis, standard care treatment as per investigator's discretion or no treatment during the next 8 weeks of the OL phase. Total duration of treatment will be of 14 weeks. Efficacy will primarily be evaluated by percentage of participants who show response as per Mayo DAI Score at Week 6. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 18 years old or older
* Participants with total Mayo DAI score between 5 to 10 at Screening and participants with score of 2 or more for the rectal bleeding and for the findings of flexible proctosigmoidoscopy or colonoscopy sub-scores of the Mayo DAI
* Participants with confirmed mild to moderate active UP not extending above rectum as evidenced by flexible proctosigmoidoscopy and histopathology assessments
* Female participants of child-bearing age who have negative serum beta-human chorionic gonadotropin (β-HCG) at the time of entry into the study
* Female participants of child-bearing age who use medically acceptable form of birth control
* Participants who are smokers and non-smokers must not change their smoking habits or nicotine use during the DB treatment period
* Participants who are literate and have legal ability to sign informed consent form

Exclusion Criteria:

* Participants with other digestive diseases interfering with the measurement of any sub-score of the Mayo DAI
* Participants with known presence or suspicion of malignant disease of the digestive system or presence or history of neoplasms other than carcinoma in situ of the cervix or basal carcinoma of the skin
* Participants with clinically significant electrocardiographic abnormalities that would compromise its participation in the study
* Participants who are chronically using oral 5-aminosalicylic acid (5-ASA) at a dose greater than 4g daily, change in the oral 5-ASA dosing, or use of any form of rectal 5-ASA formulations during the 30 days prior to randomization
* Participants with significant use of corticosteroids ,immunosuppressant's or biologic response modifiers that may have a therapeutic effect on ulcerative proctitis during the 45 days before the date of consent
* Participants who use any rectally administered medicine during the 30 days prior to randomization
* Participants who have contraindication to the use of mesalamine or suppository vehicle, analgesia, flexible proctosigmoidoscopy or colonoscopy
* Participants who have blood parameters of grade 3 or higher on the common terminology criteria for adverse events (CTCAE) 5-point scale
* Participants with severe renal or hepatic impairment with parameters of grade 3 or higher on the CTCAE
* Participants with clinically significant urinary tract obstruction and history of idiopathic pancreatitis
* Participants with presence of other known clinically significant medical and/or psychological illnesses precluding participation
* Participants who participate in clinical studies other than observational studies during the 90 days before the date of the informed consent form signature
* Participants who are unable or unwilling to complete the follow-up evaluations required for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (39):
- United States (22):
  - Birmingham Gastroenterology Associates P.C., Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Desert Sun Gastroenterology, Tucson, Arizona
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Litchfield County Gastroenterology and Associates, Torrington, Connecticut
  - Clinical Research of South Florida, Boynton Beach, Florida
  - Center for Gastrointestinal Disorders, Hollywood, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Digestive Research Associates, Newnan, Georgia
  - Advanced Pain Care Clinic, Evansville, Indiana
  - Gastrointestinal Associates, Jackson, Mississippi
  - Center for Digestive & Liver Diseases Inc., Mexico, Missouri
  - South Jersey Gastroenterology, Marlton, New Jersey
  - Synergy First Medical, Brooklyn, New York
  - Research Associates of New York (RANY), New York, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - The First Clinic, Nashville, Tennessee
  - South Texas Research Alliance, Laredo, Texas
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (8):
  - Gastroenterology & Hepatology Clinic, Abbotsford, British Columbia
  - Diamond Health Care Centre, Vancouver, British Columbia
  - Surrey GI Clinic Research, Guelph, Ontario
  - St-Joseph's Healthcare Hamilton, Hamilton, Ontario
  - DHC Research, Richmond Hill, Ontario
  - Toronto Digestive Disease Associates Inc. (TDDA), Vaughan, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
- Poland (9):
  - GASTROMED s.c., Bialystok
  - Wojewódzki Szpital Specjalistyczny Oddz. Gastroenterologii, Częstochowa
  - SPZOZ Uniwersytecki Szpital Kliniczny, Lodz
  - Wojewodzki Szpital Specjalistyczny, Lublin
  - SP Szpital Kliniczny, Lublin
  - Szpital Kolejowy, Pruszków
  - MEDICOR - Centrum Medyczne, Rzeszów
  - Endoskopia SP. Z o.o., Sopot
  - Gabinet Lekarski LECHMED, Warsaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of a total 119 double-blind phase participants, 116 participants (including 9 of the 11 participants that terminated early) further continued in the open-label (OL) phase where, under the amended protocol versions 3 and 4, they were provided the opportunity to voluntarily receive MAX-002, standard care treatment, or no treatment
Groups:
- MAX-002 (Double-blind Phase): MAX-002 suppository 1 gram (g) rectally once daily at bedtime for 6 weeks during the DB phase. Participants then received either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
- Canasa® (Double-blind Phase): Canasa® suppository 1 g rectally once daily at bedtime for 6 weeks during the DB phase. Participants then received either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
- Placebo (Double-blind Phase): Matching placebo suppository rectally once daily at bedtime, for 6 weeks during the DB phase. Participants then received either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
- MAX-002 (Open-label Phase): Participants who completed or discontinued DB phase and provided consent, received MAX-002 suppository 1 g once daily at bedtime for 8 weeks during the OL phase.
- Standard Care Treatment (Open-label Phase): Participants who completed or discontinued the DB phase and provided consent, received standard care treatment once daily for 8 weeks as per investigator's judgment during the OL phase.
- No Treatment (Open-label Phase): Participants who completed or discontinued the DB phase and provided consent, received no treatment for 8 weeks as per investigator's judgment during OL phase.
Period: Double-blind Phase
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase) | MAX-002 (Open-label Phase) | Standard Care Treatment (Open-label Phase) | No Treatment (Open-label Phase)
Started | 41 | 39 | 39 | 0 | 0 | 0
Completed | 40 | 38 | 30 | 0 | 0 | 0
Not Completed | 1 | 1 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 5 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 0 | 0 | 1 | 0 | 0 | 0
Period: Open-Label Phase
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase) | MAX-002 (Open-label Phase) | Standard Care Treatment (Open-label Phase) | No Treatment (Open-label Phase)
Started | 0 | 0 | 0 | 44 | 52 | 20
Completed | 0 | 0 | 0 | 42 | 50 | 20
Not Completed | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of Informed Consent | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Placebo (Double-blind Phase): Matching placebo suppository rectally once daily at bedtime for 6 weeks during the DB phase. Participants then received either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase
- Total: Total of all reporting groups
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase) | Total
Number analyzed (Participants) | 41 | 39 | 39 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.55) | 44.8 (11.70) | 41.8 (12.84) | 43.7 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 23 | 61
  Male | 22 | 20 | 16 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Responders at Week 6
Description: Participants were considered as responders if they had total Mayo Disease Activity Index (DAI) score less than 3 points and no individual sub-scores greater than or equal to 2. Mayo DAI is a semi-quantitative scale which consists of 4 sub-scales: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy or colonoscopy and physician global assessment, each sub-scale ranged from 0 to 3 (0=normal, 3=severe). The total Mayo DAI score ranges from 0 (normal or inactive disease) to 12 (severe disease).
Time Frame: Week 6
Population: ITT population included all randomized participants. Missing values were imputed using non-responder (NR) imputation method.
Measure: Number; unit: percentage of participants
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 41 | 39 | 39
percentage of participants | 56.1 | 46.2 | 23.1
Statistical Analysis 1: Comparison: MAX-002 (Double-blind Phase) vs Placebo (Double-blind Phase); The comparison between MAX-002 and placebo during the DB phase with respect to the primary outcome measure was the single pre-specified primary analysis, and the null hypothesis was that the percentages were equal between the two groups; Test type: Superiority or Other; p = 0.0047, Cochran-Mantel-Haenszel — Statistical significance was assessed at the two-sided 5% level. As there was only a single pre-specified primary analysis, there was no adjustment for multiplicity
Statistical Analysis 2: Comparison: Canasa® (Double-blind Phase) vs Placebo (Double-blind Phase); The comparison between Canasa® and placebo during the DB phase with respect to the primary outcome measure was a pre-specified tertiary analysis only; Test type: Superiority or Other; p = 0.0346, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Who Were Responders at Week 3
Description: Participants considered as responders if they had total Mayo DAI score less than 3 points and no individual sub-scores greater than or equal to 2. Mayo DAI is a semi-quantitative scale which consists of 4 sub-scales: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy or colonoscopy and physician global assessment, each sub-scale ranged from 0 to 3 (0=normal, 3=severe). The total Mayo DAI score ranges from 0 (normal or inactive disease) to 12 (severe disease).
Time Frame: Week 3
Population: ITT population included all randomized participants. Missing values were imputed using NR imputation method.
Measure: Number; unit: percentage of participants
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 41 | 39 | 39
percentage of participants | 36.6 | 38.5 | 12.8

3. Secondary Outcome: Time to Relief of Rectal Bleeding
Description: Time to relief of rectal bleeding was defined as number of days from randomization (Day 1) up to the first date of 3 consecutive days without observation of rectal bleeding during the double-blind phase.
Time Frame: Day 1 up to Week 6
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 41 | 39 | 39
days | 6 [4 to 9] | 5 [3 to 12] | 21 [7 to NA] — Upper limit of confidence interval was not calculable due to high number of participants who did not experience relief of rectal bleeding prior to completing or withdrawing from the study.

4. Secondary Outcome: Change From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 6
Description: The IBDQ is used to measure disease specific quality of life. The IBDQ consists of a self-administered 32-item questionnaire that evaluates quality of life across 4 domains of wellness: bowel symptoms (10 questions), systemic symptoms (5 questions), social symptoms (5 questions) and emotional function (12 questions). The response to each question is graded on 7-point likert scale, ranging from 1 (worst aspect) to 7 (best aspect). The total IBDQ is computed as the sum of the responses to the individual IBDQ questions. The total score ranges from 32 to 224 with higher scores indicating a better quality of life.
Time Frame: Baseline, Week 6
Population: The ITT population included all the participants randomized to study treatment. Missing values were imputed using remaining item average (RIA) imputation algorithm. Here 'n' signifies those participants who were evaluable at specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 41 | 39 | 39
units on a scale
  Baseline (n= 41, 39, 39) | 153.45 (35.03) | 153.19 (38.75) | 149.18 (32.40)
  Change at Week 6 (n= 41, 39, 31): number analyzed (Participants) | 41 | 39 | 31
  Change at Week 6 (n= 41, 39, 31) | 30.59 (28.95) | 42.42 (31.26) | 24.48 (27.29)

5. Secondary Outcome: Time to Relief of Tenesmus
Description: Time to relief of tenesmus (feeling of constantly needing to pass stools, even if the bowels are already empty) was defined as the number of days from randomization (Day 1) up to the first date of 3 consecutive days without observation of tenesmus during the double-blind phase.
Time Frame: Day 1 up to Week 6
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 41 | 39 | 39
days | 3 [1 to 4] | 2 [1 to 5] | 1 [1 to 10]

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (Week 14)
Description: Any event that started on or after the first dose of double-blind study medication up to completion of the last study visit (and procedures) at the end of the open-label phase.
  One participant was randomized to Placebo but received Canasa® and a second participant was randomized to MAX-002 but received Canasa® are reported under the Canasa® treatment group for the Safety population. These patients are reported under their randomized treatment group for the ITT/PP populations.
Groups:
- Placebo (Double-blind Phase): Matching placebo suppository rectally once daily at bedtime for 6 weeks during the DL phase. Participants then received either MAX-002 suppository, standard care treatment or no treatment (as per Investigator's judgment) for 8 weeks during the OL phase.
- MAX-002 (Open-label Phase): Participants who completed or discontinued the DB phase and provided consent, received MAX-002 suppository 1 g once daily at bedtime for 8 weeks during the OL phase.
Arm/Group | MAX-002 (Double-blind Phase) | Canasa® (Double-blind Phase) | Placebo (Double-blind Phase) | MAX-002 (Open-label Phase) | Standard Care Treatment (Open-label Phase) | No Treatment (Open-label Phase)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41 | 0/38 | 0/44 | 0/52 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/41 | 0/38 | 1/44 | 0/52 | 0/20
Other Adverse Events (participants affected / at risk) | 14/40 | 16/41 | 20/38 | 20/44 | 20/52 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAX-002 (Double-blind Phase) (N=40) | Canasa® (Double-blind Phase) (N=41) | Placebo (Double-blind Phase) (N=38) | MAX-002 (Open-label Phase) (N=44) | Standard Care Treatment (Open-label Phase) (N=52) | No Treatment (Open-label Phase) (N=20)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAX-002 (Double-blind Phase) (N=40) | Canasa® (Double-blind Phase) (N=41) | Placebo (Double-blind Phase) (N=38) | MAX-002 (Open-label Phase) (N=44) | Standard Care Treatment (Open-label Phase) (N=52) | No Treatment (Open-label Phase) (N=20)
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 4 | 3 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3 | 3 | 3 | 2
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 6 | 6 | 3 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Fear (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphangiectasia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated because of business/administrative reasons and not because of safety considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions may vary in accordance with each agreement that is negotiated with individual investigators. Sponsor will allow publication after multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and defer publication for period of time to allow Sponsor to obtain patent or other intellectual property right protection.